CLINICAL TRIAL: NCT04630041
Title: Implementation Barriers to Social Needs Screenings in Routine Emergency Care
Brief Title: Social Needs Screenings in ED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Andrea Wallace (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Andrea Wallace, Associate Professor, University of Utah
Organization: University of Utah (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 00125877
Record Dates: First submitted 2020-11-11; First posted 2020-11-16 (Actual); Last update posted 2020-11-16 (Actual); Status verified 2020-11

CONDITIONS: Social Determinants of Health
Keywords: Emergencies; Social needs
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Social Needs Assessment (Experimental): Patients in the Emergency Department will complete a social needs assessment screener that may refer them to 211 services
  Interventions: Behavioral: 211 Referral

INTERVENTIONS:
Behavioral: 211 Referral — Patients with one or more reported social need will be referred to 211 for community based services. 211 will reach out and contact patients for follow-up.

SUMMARY:
This study will determine whether existing Health Information Technology can be leveraged to 1) implement a universal, patient-centered social needs assessment and referral process during routine Emergency Department care; 2) understand whether linking social needs assessment, community based referral, and health outcomes data may facilitate an understanding of population health; and 3) address the needs and wishes of patients and clinicians.

Hypothesis: Results of this study will provide much needed information to already overburdened hospital systems regarding whether systematically incorporating social needs information and referrals into emergency discharge processes allows for a better understanding of factors placing patients at risk for poor outcomes post-discharge, and whether doing so has potential for enhancing discharge support for a larger patient population seen in emergency departments.

ELIGIBILITY:
Inclusion Criteria:

* seen in the UHealth University hospital ED
* ability to use touchpad technology
* ability to communicate via telephone for 211 follow-up

Exclusion Criteria:

* Non-English and non-Spanish speaking (English nor Spanish need not be the 1st language)
* unable to communicate verbally
* admitted to an inpatient unit or to a skilled nursing facility (vs discharged to a community-based setting where participants are responsible for their own self-care)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5081 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Health Utilization Outcome questionnaire | 60 days
  The variable will be created by combining primary care utilization (yes/no), ED revisit (yes/no), and hospitalization (yes/no) within 60 days of original ED visit. Scores range from 0 to 3. Higher scores indicate worse health utilization outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wallace AS, Luther BL, Sisler SM, Wong B, Guo JW. Integrating social determinants of health screening and referral during routine emergency department care: evaluation of reach and implementation challenges. Implement Sci Commun. 2021 Oct 7;2(1):114. doi: 10.1186/s43058-021-00212-y. PMID 34620248